CLINICAL TRIAL: NCT06092255
Title: A Prospective Phase I/II Clinical Study of SVZ Irradiation With Postoperative Radiotherapy in Patients With GBM.
Brief Title: A Study of SVZ Irradiation With Postoperative Radiotherapy in Patients With GBM.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Lijun Wang, Jiangsu Cancer Institute & Hospital, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZGBMRT001
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: GBM

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preventive radiotherapy irradiation SVZ group (Experimental): GBM patients who met the inclusion criteria received radiotherapy range and dose based on the EORTC outline principles. The ipsilateral and contralateral SVZ areas received 56Gy and 40Gy respectively, with a fractionated dose of 2Gy. Concurrent chemotherapy with temozolomide and six cycles of adjuvant temozolomide chemotherapy were performed at the same time as radiotherapy.
  Interventions: Radiation: Postoperative radiotherapy for SVZ

INTERVENTIONS:
Radiation: Postoperative radiotherapy for SVZ — GBM patients who met the inclusion criteria received radiotherapy range and dose based on the EORTC outline principles. The ipsilateral and contralateral SVZ areas received 56Gy and 40Gy respectively, with a fractionated dose of 2Gy. Concurrent chemotherapy with temozolomide and six cycles of adjuvant temozolomide chemotherapy were performed at the same time as radiotherapy.

SUMMARY:
This phase I/II clinical trial is intended to investigate the efficacy and safety of SVZ irradiation with postoperative radiotherapy in patients with GBM.

DETAILED DESCRIPTION:
This study is a single-center, single-arm, phase I/II clinical study. It is intended to include treatment-naïve patients with histologically or cytologically confirmed glioblastoma who have received only radical surgical treatment according to the investigator's assessment. After signing the informed consent, the patient will be selected to meet the inclusion criteria and will receive postoperative adjuvant radiotherapy combined with temozolomide chemotherapy, followed by 6 cycles of temozolomide maintenance therapy. During the follow-up process, patients included in the study can withdraw from this study if they are judged by MRI examination to have disease progression, unacceptable toxic reactions occur, or the subject decides to withdraw from the study. The subsequent specific treatment plan will be discussed with the MDT and fully discussed with the patient and family members. Implement after communication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily join this study, have the ability to understand and are willing to sign the informed consent form.

2. Aged between 18-70 years old (inclusive). 3. Newly diagnosed glioblastoma confirmed by pathology. 4. The patient must have undergone maximum surgical resection and start radiotherapy within 12 weeks after surgery.

5. MRI shows that the patient's SVZ area is involved or the distance between the tumor and the SVZ area is less than or equal to 1cm.

6. No previous brain irradiation. 7. Women of childbearing age have a negative urine test or serum pregnancy test and are contraceptive during the treatment period.

8. The ECOG performance status assessed within 7 days before the study intervention is 0-1 points.

9. Have sufficient organ function, and the subject needs to meet the following laboratory indicators:

1. Absolute neutrophil count (ANC) ≥1.5x109/L without using granulocyte colony-stimulating factor in the past 14 days.
2. Without blood transfusion in the past 14 days, platelets are ≥80×109/L.
3. Without blood transfusion or erythropoietin use in the past 14 days, hemoglobin ≥9g/dL (90g/L) or ≥5.6mmol/L.
4. Total bilirubin ≤1.5×upper limit of normal (ULN); or total bilirubin >1.5×ULN but direct bilirubin ≤SULN.
5. aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN, or subjects with liver metastasis ≤5× ULN.
6. Serum creatinine ≤ 1.5 × ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60 ml/min.
7. Good coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; or the subject is receiving anticoagulant therapy but the prothrombin time (PT) or partial thromboplastin time (PTT) is within the therapeutic range for the anticoagulant's intended use; • Activated partial thromboplastin time (aPTT) ) or partial thromboplastin time (PTT) ≤1.5 times ULN; or the subject is receiving anticoagulant therapy, but the prothrombin time (PT) or activated partial thromboplastin time (PTT) is below the expected use of the anticoagulant Within the therapeutic range;
8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, subjects can also be enrolled if total T3 (or FT3) and FT4 are within the normal range.
9. myocardial enzyme spectrum is within the normal range (such as a simple experiment that is not clinically significant in the comprehensive judgment of the researcher). Ventricular abnormalities are also allowed to be included); simple laboratory abnormalities are also allowed to be included).

Exclusion Criteria:

1. Have a personal history of malignant tumors within two years.
2. Use anti-vascular drugs such as bevacizumab before progression.
3. Women who are pregnant or breastfeeding, and women of childbearing age who are unwilling or unable to accept birth control methods during the entire study period and up to 12 weeks after the study.
4. Physical examination or clinical experimental findings that the researcher believes may interfere with the results or increase the patient's risk of treatment complications.
5. Unstable systemic accompanying diseases (active infection stage, moderate to severe chronic obstructive pulmonary disease, poorly controlled high blood pressure) Blood pressure disease, unstable angina, congestive heart failure, myocardial infarction within 6 months, severe mental disorder requiring drug control, liver, kidney or other metabolic diseases, neuropsychiatric changes such as Alzheimer's disease).
6. There may be other medical history or disease evidence that may interfere with the trial results, prevent the subject from fully participating in the study, abnormal treatment or laboratory test values, or other conditions that the researcher believes are not suitable for enrollment. The researcher believes that there are other potential risks and are not suitable for participation. this research. allowed to join the group).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 12 monnths
  Progression-free survival (PFS), defined as the time from treatment to progression or death, whichever occurs first;

SECONDARY OUTCOMES:
OS | 12 monnths
  Overall survival (OS), defined as the time from treatment to death.
Safety evaluation | 12 months
  Adverse events were assessed according to NCI CTCAE (version 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Lijun Wang, Study Director — Jiangsu Cancer Institute & Hospital
Locations (1):
- Lining Guo, Nanjing, Jiangsu, China